CLINICAL TRIAL: NCT04545515
Title: A Phase 3b Open-label Study Evaluating the Long-term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor Combination Therapy in Cystic Fibrosis Subjects Ages 6 Years and Older Who Are Heterozygous for the F508del Mutation and a Minimal Function Mutation (F/MF)
Brief Title: A Study Evaluating the Long-term Safety and Efficacy of Elexacaftor/Tezacaftor/Ivacaftor in Cystic Fibrosis (CF) Particpants 6 Years and Older and F/MF Genotypes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX20-445-119; 2020-001404-42 (EudraCT Number)
Record Dates: First submitted 2020-09-03; First posted 2020-09-11 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ELX/TEZ/IVA (Experimental): Participants 6 to less than <12 year of age and weighing <30 kilogram (kg) at Day 1 received ELX 100 milligram (mg)/TEZ 50 mg /IVA 75 mg as fixed dose combination (FDC) tablets in the morning and IVA as mono tablet in the evening and those weighing more than or equal to (≥) 30 kg at Day 1 received ELX 200 mg/TEZ 100 mg /IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 96 weeks. Doses were adjusted upward with subsequent changes in weight. Participants ≥12 years age at Day 1 received ELX 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 96 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed dose combination (FDC) tablets for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
The study evaluates the long-term safety and efficacy of elexacaftor (ELX)/tezacaftor (TEZ)/ivacaftor (IVA) triple combination (TC) in participants with CF who are 6 years of age and older with F/MF genotypes.

ELIGIBILITY:
Key Inclusion Criteria:

* Completed study drug treatment in parent study (VX19-445-116, NCT04353817), or had study drug interruption(s) in parent study but completed study visits up to the last scheduled visit of the treatment period in the parent study

Key Exclusion Criteria:

* History of study drug intolerance in the parent study

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- Australia (3):
  - Telethon Kids Institute, Nedlands
  - Queensland Children's Hospital, South Brisbane
  - The Children's Hospital at Westmead, Westmead
- Canada (3):
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Juliane Marie Center, Rigshospitalet, Copenhagen, Denmark
- France (5):
  - Groupe Hospitaler Pellegrin, CHU De Bordeaux, Bordeaux
  - CHU Lyon - Hopital Femme Mere-Enfant, Bron
  - Hopital Necker, Enfants Malades, Paris
  - Hopital Robert Debre, Paris
  - Centre de Perharidy, Roscoff
- Germany (7):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitaetsklinkum Koeln, CF-Studienzentrum, Cologne
  - Universitatsklinikum Essen (AoR), Kinderklinik III, Abt. fur Pneumologie, Essen
  - Johann Wolfgang Goethe University, Frankfurt
  - Justus-Liebig-Universität Gießen Zentrum fur Kinderheilkunde und Jugendmedizin, Giessen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Heidelberg, Zenter fuer Kinder-und Jugendmedizin, Heidelberg
- Israel (2):
  - Hadassah University Hospital Mount Scopus, Jerusalem
  - Schneider Children's Medical Center of Israel, Petach Tikvah
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medical Center / Sophia Children's Hospital, Rotterdam
- Spain (2):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Virgen de la Arrixaca, Murcia
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Kinderspital Zuerich, Zurich
- United Kingdom (7):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol Royal Hospital, Bristol
  - Children's Hospital of Wales, Cardiff
  - Royal Hospital for Sick Children, Edinburgh
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Sick Children, London
  - Royal Brompton & Harefield NHS Foundation Trust, Royal Brompton Hospital, London
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 120 participants from the parent study VX19-445-116 (NCT04353817) were enrolled in this study.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA
Started | 120
Placebo-ELX/TEZ/IVA (Participants from the Placebo group of the parent study VX19-445-116, who received ELX/TEZ/IVA during the current study VX20-445-119.) | 61
ELX/TEZ/IVA-ELX/TEZ/IVA (Participants from the ELX/TEZ/IVA group of the parent study VX19-445-116, who continued to receive ELX/TEZ/IVA during the current study VX20-445-119.) | 59
Completed | 110
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Withdrawal of consent (not due to AE) | 2
Not completed — Commercial drug is available for participant | 7

BASELINE CHARACTERISTICS:
Population: Baseline data for the long-term safety analysis is based on the parent study baseline, which is defined as the most recent non-missing measurement collected before the first dose of study drug in the treatment period of parent study.
Groups:
- ELX/TEZ/IVA: Participants 6 to <12 year of age and weighing <30 kg at Day 1 received ELX 100 mg/TEZ 50 mg /IVA 75 mg as FDC tablets in the morning and IVA as mono tablet in the evening and those weighing ≥30 kg at Day 1 received ELX 200 mg/TEZ 100 mg /IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 96 weeks. Doses were adjusted upward with subsequent changes in weight. Participants ≥12 years age at Day 1 received ELX 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 96 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 90
  Not collected per local regulations | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87
  Black or African American | 1
  Asian | 1
  American Indian or Alaska Native | 1
  Other | 1
  Not collected per local Regulations | 28
  Multiracial | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: From Baseline up to Week 100
Population: The Open-label Safety Set (OL-SS) included all participants who had received at least 1 dose of study drug in the Open label extension (OLE) study.
Measure: Count of Participants; unit: Participants
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 120
Participants
  Participants with TEAEs | 118
  Participants with SAEs | 13

2. Secondary Outcome: Absolute Change From Parent Study Baseline in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Parent Study Baseline to Week 96
Population: OL Full Analysis Set (OL-FAS) included all enrolled participants who received at least 1 dose of study drug in this study. Data were planned to be presented as per parent study reporting groups (i.e. Placebo-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA). Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome at Week 96 and "Number Analyzed" signifies participants who were evaluable in the specified parent study reporting group.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 98
millimole per liter (mmol/L)
  Placebo (Parent study)-ELX/TEZ/IVA (Current study): number analyzed (Participants) | 52
  Placebo (Parent study)-ELX/TEZ/IVA (Current study) | -57.3 (2.2)
  ELX/TEZ/IVA (Parent study)-ELX/TEZ/IVA (Current study): number analyzed (Participants) | 46
  ELX/TEZ/IVA (Parent study)-ELX/TEZ/IVA (Current study) | -57.5 (2.3)

3. Secondary Outcome: Absolute Change From Parent Study Baseline in Lung Clearance Index 2.5 (LCI2.5)
Description: The LCI2.5 index is the number of lung turnovers required to reduce the end tidal inert gas concentration to 1/40th of its starting values and is calculated by dividing the sum of exhaled tidal breaths (cumulative exhaled volume (CEV)) by simultaneously measured functional residual capacity (FRC). An LCI of 7.5 and below is normal; values greater than 7.5 are abnormal. LCI is able to detect abnormalities in lung function earlier than more traditional modalities such as spirometry.
Time Frame: From Parent Study Baseline to Week 96
Population: OL-FAS. Data were planned to be presented as per parent study reporting groups (i.e. Placebo-ELX/TEZ/IVA and ELX/TEZ/IVA-ELX/TEZ/IVA). Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome at Week 96 and "Number Analyzed" signifies participants who were evaluable in the specified parent study reporting group.
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 104
Index
  Placebo (Parent study)-ELX/TEZ/IVA (Current study): number analyzed (Participants) | 56
  Placebo (Parent study)-ELX/TEZ/IVA (Current study) | -1.74 (0.18)
  ELX/TEZ/IVA (Parent study)-ELX/TEZ/IVA (Current study): number analyzed (Participants) | 48
  ELX/TEZ/IVA (Parent study)-ELX/TEZ/IVA (Current study) | -2.35 (0.19)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 100
Description: The OL-SS included all participants who had received at least 1 dose of study drug in the OLE study.
Arm/Group | ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/120
Serious Adverse Events (participants affected / at risk) | 13/120
Other Adverse Events (participants affected / at risk) | 118/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=120)
Constipation (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Steatorrhoea (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 1
Bacterial disease carrier (Infections and infestations) | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2
Pneumonia pseudomonal (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Blood glucose increased (Investigations) | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Weight gain poor (Metabolism and nutrition disorders) | 1
Haematuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=120)
Ear pain (Ear and labyrinth disorders) | 8
Conjunctivitis allergic (Eye disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 27
Abdominal pain upper (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 24
Fatigue (General disorders) | 6
Pyrexia (General disorders) | 48
Immunisation reaction (Immune system disorders) | 8
Bacterial disease carrier (Infections and infestations) | 8
COVID-19 (Infections and infestations) | 70
Hordeolum (Infections and infestations) | 10
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 19
Influenza (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 54
Rhinitis (Infections and infestations) | 29
Upper respiratory tract infection (Infections and infestations) | 37
Viral upper respiratory tract infection (Infections and infestations) | 13
Alanine aminotransferase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 6
Bacterial test positive (Investigations) | 7
SARS-CoV-2 test positive (Investigations) | 12
Staphylococcus test positive (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Headache (Nervous system disorders) | 45
Cough (Respiratory, thoracic and mediastinal disorders) | 62
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT04545515/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT04545515/SAP_001.pdf